CLINICAL TRIAL: NCT03404479
Title: A Prospective, Randomized, Double-blinded, Multi-center, Trial to Evaluate Efficacy and Safety of Combination of Diacerein and Celecoxib Administered Orally in Patients With Knee Osteoarthritis
Brief Title: Trial to Evaluate Efficacy and Safety of Combination of Diacerein and Celecoxib Administered in Patients With Knee OA
Acronym: DIA IIT_01
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Whan-Seok Choi (Other)
Collaborators: Korea University Guro Hospital (Other)
Responsible Party: Sponsor-Investigator, Whan-Seok Choi, Professor, Seoul St. Mary's Hospital
Organization: Seoul St. Mary's Hospital (Other)
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: DIA IIT_01
Record Dates: First submitted 2018-01-12; First posted 2018-01-19 (Actual); Last update posted 2018-02-26 (Actual); Status verified 2018-02

CONDITIONS: Knee Osteoarthritis
Keywords: Knee Osteoarthritis; Diacerein
MeSH Terms: conditions — Osteoarthritis, Knee | interventions — diacerein; Celecoxib

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Co-administration group (Experimental): Co-administration of Diacerein 50mg, Celecoxib 100mg.
  Interventions: Drug: Diacerein; Drug: Celecoxib
- Single administration group 1 (Active Comparator): Single administration of Diacerein 50mg and placebo.
  Interventions: Drug: Diacerein
- Single administration group 2 (Active Comparator): Single administration of Celecoxib 100mg and placebo.
  Interventions: Drug: Celecoxib

INTERVENTIONS:
Drug: Diacerein — For 12 weeks, administered twice a day by oral.
  Arms: Co-administration group; Single administration group 1
Drug: Celecoxib — For 12 weeks, administered twice a day by oral.
  Arms: Co-administration group; Single administration group 2

SUMMARY:
The purpose of this study is to evaluate the pain relief effect of Co-administration of Diacerein with Celecoxib in patients with knee osteoarthritis compared with single administration of each drug.

DETAILED DESCRIPTION:
A large epidemiological study in Europe reported that over four-thirds of patients with osteoarthritis received combination therapy with two or more drugs. Approximately 1.5% of patients with osteoarthritis using three or more drugs are using COX-2(Cyclo-oxygenase-2) inhibitors and SYSADOA(Symptomatic slow acting drug), And it has been investigated that much more patients are using the two classes of drugs when the range is extended to other oral NSAIDs other than COX-2 inhibitors. Therefore, considering the characteristics of patients with osteoarthritis, such as basal disease and treatment effects on each type of drug, it is important to find the optimal combination of drugs for each patient characteristics.

There is a previous study using osteoarthritis rat model as a biological basis of diacerein and celecoxib administration. Previous studies have shown that the combined use of Diacerein and Celecoxib improves osteoarthritis.

The purpose of this study is to evaluate the pain relief effect of Co-administration of Diacerein with Celecoxib in patients with knee osteoarthritis compared with single administration of each drug.

ELIGIBILITY:
Inclusion Criteria:

1. Subjects who voluntarily consented, after listening enough explanation for this study and investigational product.
2. Adult over 50 years of age.
3. At least one of the knee pain VAS score is 40mm or more.
4. Meets the ACR(American College of Rheumatology) criteria for diagnosis. (1) Confirmation of osteophytes on radiographic inspection. (2) One or more of the following three items.

   ① Age> 50 years

   ② Morning stiffness <30 minutes

   ③ Crepitus
5. Patients who require medication for more than 12 weeks due to osteoarthritis symptoms.
6. Those who are able to follow the requirements of this clinical trial, such as being able to trace during the clinical trial period and to read and write the VAS questionnaire.
7. Those who weigh more than 40kg

Exclusion Criteria:

1. Secondary knee osteoarthritis
2. Other inflammatory Knee Osteoarthritis (e.g. gout, rheumatoid arthritis, etc.)
3. Patients presenting with gastroesophageal reflux disease, peptic ulcer.
4. Helicobacter infected patients who have not been treated for eradication (recruitment if negative in re-examination after treatment).
5. Short bowel syndrome that can cause inflammatory bowel disease (ulcerative colitis, Crohn's disease) and drug absorption disorder.
6. Intestinal obstruction syndrome
7. Unexplained abdominal pain
8. ALT(Alanine aminotransferase) level of liver function test exceeded 5 times of reference range
9. Total bilirubin level exceeded 2 mg / dL
10. Serum albumin level less than 2 g / dL
11. Ascites
12. Hepatic encephalopathy
13. Hepatitis B, hepatitis C (excluding healthy carriers) or HIV positive
14. MDRD(Modification of Diet in Renal Disease) Estimated Glomerular filtration rate less than 60 mL / m2
15. Patients with hyperkalemia (over 5.5 meq / L)
16. history of asthma, acute rhinitis, nasal polyps, angioedema, urticaria or allergic reactions to aspirin or other non-steroidal anti-inflammatory drugs(including COX-2 inhibitors).
17. Malignant tumors other than basal cell or squamous cell carcinoma of the skin, CIN(Cervical Intraepitherial Neoplasia) and CIS(Carcinoma in situ) of the cervix, and intraepithelial carcinoma of other areas Within 5 years of consent date.
18. Medical history of hypersensitivity to the components of the investigational products. (The components of test drug 1 and 2, including the Rhein-based drug)
19. Patients with an allergic reaction to sulfonamide.
20. Patients with galactose intolerance, lapp lactase deficiency or glucose-galactose malabsorption.
21. Subjects who have not reached the prescribed period after receiving contraindicated medication or treatment before participation in this clinical trial.
22. Patients receiving contraindicated medication.
23. Alcohol and other drug abuse cases based on 6 months before screening.
24. Pregnant women or nursing mothers who are not willing to stop breastfeeding.
25. Female who do not fall into one or more of the following categories(In other words, only the following female can participate:)

    * (1) Menopause (non-therapy-induced amenorrhea of more than 12 months) Female
    * (2) Female infertility due to surgery (no ovaries and / or uterus)
    * (3) If you have sexual intercourse with only one male partner who has been confirmed to have no semen after fertilization.
    * (4) Female subjects who agreed to abstinence during the clinical trial period.
    * If the subject is assured of an abstinence throughout the trial period.(e.g. clergy)
    * However, intermittent abstinence (eg, contraception using ovulation period, symptothermal) or coitus interrupts is not a case of consent for abstinence.
    * (5) For women of childbearing age, the following methods or methods of contraception use the effective method of contraception to be used during the period of this clinical trial:
    * Oral contraceptive
    * The contraceptive patch
    * Intra uterine device (IUD)
    * contraceptive implant
    * contraceptive injection
    * intrauterine hormonal apparatus
    * Tubal ligation and infertility surgery
26. If 30 days have not elapsed after the date of signing of the previous clinical trial or currently participating in other clinical trials.
27. Patients who are scheduled for surgery during the clinical trial period or who have difficulties in completing the protocol during this clinical trial due to other reasons.
28. In addition to the above, other diseases that the investigator judges to be inappropriate.

Min Age: 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 90 (Estimated)
Dates: Start 2018-01-25 (Actual); Primary Completion 2019-01-02 (Estimated); Study Completion 2019-01-02 (Estimated)

PRIMARY OUTCOMES:
pain VAS score | 12 weeks after randomization
  Changes in pain VAS(Visual analogue scale) score before and after 12 weeks of drugs administration.
  (No pain score: 0, Worst pain score: 100)

SECONDARY OUTCOMES:
pain NRS score | 12 weeks after randomization
  Changes in pain NRS(Numeric rating scale) score before and after 12 weeks of drugs administration.
  (No pain score: 0, Worst pain score: 10)
WOMAC index score | 12 weeks after randomization
  Changes in WOMAC(Western Ontario and mcmaster Universities Osteoarthritis Index) index score before and after 12 weeks of drugs administration (possible score range, Pain: 0-20, Stiffness: 0-8, Physical function: 0-68; Total Score range: 0-96 ('none' to 'extreme'))
GSRS index score | 12 weeks after randomization
  Changes in GSRS(Gastrointestinal symptom rating scale) index score before and after 12 weeks of drugs administration.
  (Score range: 0-45 ('none' to 'extreme'))

CONTACTS AND LOCATIONS:
Overall Officials: Whan-Seok Choi, MD, PhD, Principal Investigator — Seoul St. Mary's Hospital; Seon-Mee Kim, MD, PhD, Principal Investigator — Korea University Guro Hospital
Locations (2):
- South Korea (2):
  - Seoul ST. Mary's Hospital, Seoul
  - Korea University Guro Hospital, Seoul

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Li Z, Meng D, Li G, Xu J, Tian K, Li Y. Celecoxib Combined with Diacerein Effectively Alleviates Osteoarthritis in Rats via Regulating JNK and p38MAPK Signaling Pathways. Inflammation. 2015 Aug;38(4):1563-72. doi: 10.1007/s10753-015-0131-3. PMID 25687638
- [Background] Martel-Pelletier J, Pelletier JP. Effects of diacerein at the molecular level in the osteoarthritis disease process. Ther Adv Musculoskelet Dis. 2010 Apr;2(2):95-104. doi: 10.1177/1759720X09359104. PMID 22870441
- [Background] Panova E, Jones G. Benefit-risk assessment of diacerein in the treatment of osteoarthritis. Drug Saf. 2015 Mar;38(3):245-52. doi: 10.1007/s40264-015-0266-z. PMID 25652235
- [Background] Nicolas P, Tod M, Padoin C, Petitjean O. Clinical pharmacokinetics of diacerein. Clin Pharmacokinet. 1998 Nov;35(5):347-59. doi: 10.2165/00003088-199835050-00002. PMID 9839088